CLINICAL TRIAL: NCT03961568
Title: A Multicenter Open-Label Extension Study to Evaluate the Long-Term Safety of Cenobamate Adjunctive Therapy in Subjects With Primary Generalized Tonic-Clonic Seizures
Brief Title: Cenobamate Open-Label Extension Study for YKP3089C025
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YKP3089C033
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Primary Generalized Tonic Clonic Seizures in the Setting of Idiopathic Generalized Epilepsy
Keywords: Idiopathic Generalized Epilepsy
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized | interventions — Cenobamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Core Study Placebo (Experimental): Subjects who did not receive Cenobamate in the Core Study will receive Cenobamate 12.5 mg tablet once a day for two weeks, 25 mg tablet once a day for two weeks, 50 mg tablet once a day for two weeks, 100 mg tablets once a day for two weeks, 150 mg tablets once a day for two weeks and 200 mg tablets once a day for twelve weeks.
  Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight.
  Interventions: Drug: Cenobamate
- Core Study Active (Experimental): Subjects who received cenobamate in the Core study will continue to receive the same daily dose (150 mg or 200mg).
  Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight.
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — active drug
  Other Names: YKP3089

SUMMARY:
52 Week Open-Label Safety Study of Cenobamate for Subjects who Complete YKP3089C025 (core study)

DETAILED DESCRIPTION:
52 Week Open-Label Safety Study of cenobamate adjunctive therapy for subjects who complete double-blind study YKP3089C025. Subjects will have a 12 week double-blind conversion phase where subjects who received placebo in the double-blind study will be converted to cenobamate. Subjects who received cenobamate in the double-blind study will continue to receive their daily dose of cenobamate. Subjects switching from placebo to cenobamate will be titrated starting at 12.5 mg and increase their dose over the course of 12 weeks as follows 12.5 mg for 2 weeks, 25 mg for two weeks, 50 mg for two weeks, 100 mg for two weeks, 150 mg for two weeks, and 200 mg for two weeks. All subjects will receive 200 mg for the last two weeks of the conversion phase to preserve the blind. After completing the double-blind conversion phase, subjects will have 40 weeks of open-label, flexibly dosed cenobamate. The dose range is 50 mg - 200 mg. Primary endpoints are all safety measures.

Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight

ELIGIBILITY:
Inclusion Criteria:

* The subject must have successfully completed the Double-blind Treatment Period in the Core study.
* Written informed consent signed by the subject or legal guardian, prior to entering the study, in accordance with the International Council for Harmonisation (ICH) Good Clinical Practice (GCP) guidelines. If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained. As required by country-specific regulations, only the subject may sign the ICF in accordance with ICH guidelines.

Exclusion Criteria:

* Subject tests positive, via urine drug screen at Visit 14 of the Core study, for illicit drugs except for tetrahydrocannabinol and Cannabinoids.
* Any significant changes to the subject's medical history that, in the opinion of the Principal Investigator, could affect the subject's safety or conduct of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and SAEs | 386 +/- 2 days
  Summary statistics for clinical laboratory test results and vital signs; and physical examination, neurologic examination and electrocardiogram (ECG) finding.

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Misra, MD, Study Director — SK Life Science, Inc.
Locations (45):
- United States (16):
  - University of California, San Diego (UCSD), La Jolla, California
  - The Neurology Research Group, LLC., Miami, Florida
  - University of South Florida, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Maine Medical Center, Scarborough, Maine
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Missouri Medical School, Columbia, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Five Towns Neuroscience Research, Woodmere, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Valley Medical Center, Renton, Washington
  - MultiCare Rockwood Neurology Center, Spokane, Washington
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Diagnostic Consultative Center Neoclinic EAD, Sofia
  - Diagnostic Consultative Center Equita EOOD, Varna
  - Medical Center Medica Plus OOD, Veliko Tarnovo
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski Gorna Oryahovitsa EOOD, Veliko Tarnovo
- Czechia (4):
  - Cerebrovaskularni poradna, Ostrava-Poruba
  - Fakultni nemocnice v Motole, Prague
  - Forbeli s.r.o.-Neurologicka ambulance, Prague
  - Neurologicka ambulance, Zlín
- Semmelweis Egyetem I. Sz. Gyermekgyogyaszati Klinika, Budapest, Hungary
- Poland (4):
  - Clinical Research Center Spólka z Ograniczona Odpowiedzialnoscia Medic-R sp. k., Poznan, Greater Poland Voivodeship
  - Centrum Leczenia Padaczki i Migreny, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Pratia Warszawa, Warsaw, Masovian Voivodeship
  - Górnoslaskie Centrum Medyczne im. prof. Leszka Gieca Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
- Slovakia (3):
  - MUDr. Beata Dupejova, neurologicka ambulancia, s.r.o., Banská Bystrica
  - IN MEDIC s.r.o., Bardejov
  - Konzilium, s.r.o., Dubnica nad Váhom
- Ukraine (11):
  - Municipal Institution "Dnipropetrovsk City Clinical Hospital No16" of Dnipropetrovsk Regional Council, Dnipro, Dnipropetrovsk Oblast
  - Municipal Institution Odesa Regional Clinical Hospital, Department of Cerebro-Vascular Diseases, Odesa, Odesa Oblast
  - Regional Clinical Center of Neurosurgery and Neurology "Uzhhorod National University", Uzhhorod, Zakarpattia Oblast
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhya, Zaporizhzhya
  - Communal Institution "Dnipropetrovsk Regional Clinical Hospital n.a. I.I. Mechnikov", Regional Center, Dnipro
  - Municipal Institution "Dnipropetrovsk Regional Clinical Hospital named after I. I. Mechnikov", Dnipro
  - Regional Psyconeurology Hospital #3, Ivano-Frankivsk
  - Communal Non-Commercial Enterprise of Kharkiv Regional Council, Kharkiv
  - Municipal Institution of Lviv Regional Council, Lviv
  - Ternopil Regional Municipal Psychoneurological Hospital, Ternopil
  - Municipal Institution "Vinnytsia Regional Psychoneurological Hospital named after Acad. O.I. Yushch, Vinnytsia